CLINICAL TRIAL: NCT04430218
Title: Peripheral Interfaces in Amputees for Sensorimotor Integration
Acronym: iSens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency); Case Western Reserve University (Other); University Hospitals Cleveland Medical Center (Other); MetroHealth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: A3355-R; RX003355-01 (Other Grant/Funding Number: VA RR&D); HT94252510204 (Other Grant/Funding Number: Department of Defense (CDMRP)); 1612632 (Other: IRBnet); CDMRP-PR241366 (Other: CDMRP-eBRAP Log number)
Record Dates: First submitted 2020-05-12; First posted 2020-06-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Upper Extremity Amputee
Keywords: Sensory Feedback; Advanced Control; Sensorimotor feedback; Prostheses and implants

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized clinical trial in a small population of subjects to answer the primary question of whether use of a sensory-enabled, high degree-of-freedom (SE-ihDOF) prosthesis with the iSens system improves the subject's quality of life compared to use of their prescribed state-of-art (SOA) prosthesis
Who Masked: Outcomes Assessor
Masking Description: The assessments will be analyzed by a blinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- iSens (Experimental): 3 months trial with the iSens system
  Interventions: Device: iSens
- State of the Art Prosthesis (No Intervention): 3 months trial with their own prosthesis.

INTERVENTIONS:
Device: iSens — The study involves a surgical implant of cuff electrodes on the nerves in the amputated limb, and muscle recording electrodes the remaining muscles. These will be connected to an implanted stimulator. The stimulator will connect wirelessly to an advanced prosthesis. This may allow a user to move the prosthetic hand intuitively and feel what your prosthesis is touching.
  Arms: iSens

SUMMARY:
The purpose of this research is to gather information on the safety and effectiveness of an implanted wireless sensory enabled highly intuitive controlled prosthetic device.

DETAILED DESCRIPTION:
The study involves a surgical implant of cuff electrodes on the residual nerves in the amputated limb, and muscle recording electrodes in muscles. These will be connected to an implanted stimulator. The stimulator will connect wirelessly to an advanced prosthesis. This may allow the user to move the prosthetic hand intuitively and feel what the prosthesis is touching.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or greater
* Acquired upper limb amputation
* Unilateral or bilateral amputation, Above or below elbow
* At least 6 months since time of amputation
* Current user of a myoelectric prosthesis or prescribed to use one
* Viable target nerves in the upper extremity *
* Recommendation from a psychologist following a psychological assessment that the subject is mentally competent and capable of completing the study related activities

Exclusion Criteria:

* A contraindication preventing surgery
* Uncontrolled diabetes
* Chronic skin ulcerations
* History of poor wound healing without specific cause
* History of uncontrolled infection without specific cause
* Active infection
* Pregnancy or women of childbearing potential unwilling to prevent pregnancy during participation in the study
* Inability to speak English
* Expectation that MRI will be required at any point for duration of study or while device is implanted.
* Arthritis in the area of implant
* Individuals with active implantable medical devices or individuals that use external active medical devices that are medically necessary and/or life-supporting or life-sustaining (e.g. insulin pumps, ventilators)
* Presence of auto immune diseases, or conditions requiring immunosuppression.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Experience Measure | 9 months post implant
  Consists of 49 items and consists of five subscales, measuring Self-efficacy, Embodiment, Body image, Prosthesis Efficiency, and Social Touch. Each scale is scored individually, and a higher score indicates a better outcome.

SECONDARY OUTCOMES:
Modified Box and Blocks | 9 months post implant
  Measuring the change in numbers of blocks moved during a timed test.

CONTACTS AND LOCATIONS:
Overall Officials: Emily L Graczyk, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (2):
- United States (2):
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Case Western Reserve University, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be uploaded to a data repository.

REFERENCES:
- [Derived] Cady SR, Lambrecht J, Tyler DJ. Enhanced sensory perception and myoelectric control with high channel count implanted sensorimotor systems. J Neural Eng. 2025 Dec 9;22(6):066024. doi: 10.1088/1741-2552/ae24ae. PMID 41297066
- [Derived] Cady SR, Lambrecht JM, Dsouza KT, Dunning JL, Anderson JR, Malone KJ, Chepla KJ, Graczyk EL, Tyler DJ. First-in-human implementation of a bidirectional somatosensory neuroprosthetic system with wireless communication. J Neuroeng Rehabil. 2025 Apr 23;22(1):90. doi: 10.1186/s12984-025-01613-z. PMID 40269935
- [Derived] Lambrecht JM, Cady SR, Peterson EJ, Dunning JL, Dinsmoor DA, Pape F, Graczyk EL, Tyler DJ. A distributed, high-channel-count, implanted bidirectional system for restoration of somatosensation and myoelectric control. J Neural Eng. 2024 Jun 21;21(3). doi: 10.1088/1741-2552/ad56c9. PMID 38861967